CLINICAL TRIAL: NCT01707615
Title: Beneficial Effects of Grape Seed Proanthocyanidin Extrat on Progression of Carotid Intima-media Thickness and Atherosclerotic Plaques in Clinical Use
Brief Title: Beneficial Effects of Grape Seed Proanthocyanidin Extrat on Progression of Atherosclerotic Plaques in Clinical Use
Acronym: GSPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jie Qiu (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Jie Qiu, Qilu Hospital of Shandong University, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010GGC10294
Record Dates: First submitted 2012-08-14; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Atherosclerosis of Arteries of the Extremities, Unspecified
Keywords: proanthocyanidin,atherosclerosis, carotid plaque
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Other): In the control group, all patients were enrolled in a lifestyle intervention
  Interventions: Other: lifestyle intervention
- GSPE group (Active Comparator): GSPE 240 mg/day (120mg bid) in addition to the same lifestyle intervention.
  Interventions: Drug: GSPE; Other: lifestyle intervention

INTERVENTIONS:
Drug: GSPE — GSPE 240 mg/day (120mg bid)
  Other Names: Grape seed proanthocyanidin extrat
  Arms: GSPE group
Other: lifestyle intervention — dietary modification making the total ingestion of calories into standard body weight 25 kCal in effect and an individualized home exercise program of a minimum 150 min/week of moderate-intensity physical activity

SUMMARY:
The purpose of this study is to investigate the antiatherogenic effect of GSPE in clinical use

DETAILED DESCRIPTION:
Atherosclerotic plaques indicate the occurrence of ischemia events and how to deal with it is a difficult task for clinical physicians. Grape seed proanthocyanidin extrat (GSPE) has been reported to exert an antiatherogenic effect by inducing regression of atherosclerotic plaques in animal experimental studies. In this study, the antiatherogenic effect of GSPE has been investigated in clinical use.

ELIGIBILITY:
Inclusion Criteria:

* (1) carotid ultrasound examination: presence of carotid plaque or abnormal CIMT of between 0.9 and 1.2mm; (2) lipid profile: LDL≦3.12mmol/L, TC≦5.2mmol/L; (3) no lipid-lowering treatment within the past 6 months.

Exclusion Criteria:

* severe cardiomyopathy, acute coronary syndrome, hepatic dysfunction, end-stage renal failure (serum creatinine ≥117mmol/L), prior carotid endarterectomy, and/or patients who did not agree to participate in the present study.

Ages: 43 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Carotid B-Mode Ultrasound | Carotid ultrasound examination was performed at baseline and 6, 12, 24months after treatment.The change of carotid plaque was record within 24 months.
  The common, internal, and external carotid arteries were carefully identified by combining B-mode ultrasonography and color-Doppler duplex examination in the anterior oblique, lateral, and posterior oblique planes. All data was collected in 12 segments: the near （intimal-luminal surface) and far (medial- adventitial) walls of the distal common (1 cm proximal to dilation of the carotid bulb), the bifurcation (1cm proximal to the flow divider), and the proximal internal (1 cm section of the internal carotid artery immediately distal to the flow divider) left and right carotid artery.

SECONDARY OUTCOMES:
clinical vascular events | after 24 months follow-up
  including hospital readmission for unstable angina, myocardial infarction, stroke, TIA, an arterial revascularization procedure (percutaneous coronary revascularization or coronary bypass surgery) and cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiu, doctor, Study Director — Qilu Hospital of Shandong University